CLINICAL TRIAL: NCT03396666
Title: Impact of a Mobile Tele-rehabilitation Solution on Body Composition of Obese Patients.
Brief Title: Mobile Tele-rehabilitation Solution for Obese Patients.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inclusion of the last Patient
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL17_0031; 2017-A01190-53 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2021-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telemouv (Experimental): Telemouv telerehabilitation solution Patients will receive telerehabilitation solution during three months
  Interventions: Other: Telemouv
- No intervention (No Intervention): Regular follow-up with advice on physical activity and nutrition

INTERVENTIONS:
Other: Telemouv — Telemouv telerehabilitation solution Patients will receive telerehabilitation solution during three months
  Arms: Telemouv

SUMMARY:
Published data indicate that rehabilitation in obese patients can result in a loss of body fat and weight that is correlated to improved physical and psychological condition and reduced morbidity and mortality.

the Ivestigators hypothezise that the use of a mobile telerehabilitation solution will encourage the patient to adopt behavioral modifications allowing a reduction of fat mass

DETAILED DESCRIPTION:
Obesity is one of the most important public health care problems worldwide and is associated with increased morbidity and mortality and high healthcare costs. Not all obese patients have the same metabolic risk. It is pejorated in case of increase in the fat mass (FM) and especially when it predominates at the visceral abdominal level.

Clinical trials have established the efficacy of lifestyle and behavioral interventions in obesity.

The recent development of telerehabilitation is a promising approach that has only been the subject of pilot studies Therefore, the investigators aim to test the effects of 3 months of telerehabilitation solution on fat mass evaluated by impedance analysis.

The telerehabilitation program Telemouv includes physical activity sessions with low intensity endurance training targeted at the level of maximal oxidation, nutritional monitoring, therapeutic education tools and motivational support

Patients with BMI > 30 kg/m² will be randomized for the intervention.

The investigators also will analyse the effects of the solution on different anthropometric, metabolic,cardiovascular and psychological parameters, and on rest and exercise metabolism. Moreover, we will assess behavioural changes in physical activity and nutrition

At the end of the study, patients in the control group will be able to benefit from the telemouv solution in an ancillary study with a follow-up of three months.

For a alpha threshold of 5% and a study power of 90%, the study should include 22 patients in each group. Taking in account a possible 10% of dropout the study will need to include 25 patients by randomized arm to demonstrate an effect.

ELIGIBILITY:
Inclusion criteria:

* Body Mass Index > 30 kg/m²
* Age 20-65 years

Exclusion criteria:

* Unstabilized primary pathologies (cardiovascular, renal, metabolic, psychiatric)
* No internet access at home

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Modification of the amount of fat mass | Month 3
  Modification of the amount of fat mass, expressed in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bughin F, Bui G, Ayoub B, Blervaque L, Saey D, Avignon A, Brun JF, Molinari N, Pomies P, Mercier J, Gouzi F, Hayot M. Impact of a Mobile Telerehabilitation Solution on Metabolic Health Outcomes and Rehabilitation Adherence in Patients With Obesity: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Dec 6;9(12):e28242. doi: 10.2196/28242. PMID 34874887